CLINICAL TRIAL: NCT00225576
Title: Statewide Implementation of Electronic Health Records
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Collaborators: Massachusetts eHealth Collaborative (Other)
Responsible Party: Principal Investigator, david bates, Chief of General Medicine, BWH, Agency for Healthcare Research and Quality (AHRQ)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HS015397
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Medication Errors
Keywords: medication errors; adverse drug events; electronic health records
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Paper prescribing, 2005 and 2007
- 2 (Experimental): Paper prescribing 2005 vs. electronic prescribing 2007
  Interventions: Other: Electronic Health Record Implementation

INTERVENTIONS:
Other: Electronic Health Record Implementation — Intervention subjects implemented electronic prescribing as part of an electronic health record implementation
  Other Names: eClinical Works
  Arms: 2

SUMMARY:
To determine the effects of Electronic Health Record use on medication error rates in primary care office practices.

Hypothesis: Adoption of Electronic Health Records through this program will reduce medication errors

DETAILED DESCRIPTION:
From the practices committed to implementing EHR in early 2005, we randomly selected 15 adult community-based primary care physicians. We selected 15 similar physicians in practices that were not planning to adopt in that time period.

At each of these physicians' practices we documented rates of medication errors for one week prior to the implementation of an EHR using duplicate prescription pads. Two months after the implementation in the adopting group, allowing some time for familiarization with the tool, we collected two weeks of data using computer-based information (in the adopting arm) and duplicate prescriptions (in the non-adopting arm).

ELIGIBILITY:
Inclusion Criteria:

* All patients of physicians participating in the study

Exclusion Criteria:

* Any patients who are not part of a panel of a participating physician
* Any patients who are younger than 18 years of age
* Any patients who came in for a second visit within each data collection period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2030 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
1. Medication errors | 2005-2007
2. Near misses | 2005-2007
3. Adverse drug events | 2005-2007

CONTACTS AND LOCATIONS:
Overall Officials: David W. Bates, MD, MPH, Principal Investigator — Brigham and Women's Hospital, Partners Healthcare System Inc.; Rainu Kaushal, MD, MPH, Principal Investigator — Cornell Weill Medical College
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Abramson EL, Bates DW, Jenter C, Volk LA, Barron Y, Quaresimo J, Seger AC, Burdick E, Simon S, Kaushal R. Ambulatory prescribing errors among community-based providers in two states. J Am Med Inform Assoc. 2012 Jul-Aug;19(4):644-8. doi: 10.1136/amiajnl-2011-000345. Epub 2011 Dec 1. PMID 22140209